CLINICAL TRIAL: NCT01665716
Title: Ovarian Ageing in Type 1 Diabetes Mellitus: the Role of Vascular Factors
Brief Title: Ovarian Ageing in Type 1 Diabetes Mellitus
Acronym: OVADIA
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Frank JM Broekmans, Prof. Dr. F. J. M. Broekmans, UMC Utrecht
Other Study IDs: NL32242.041.10; 10-345 (Other: Medical Ethics Committee UMC Utrecht)
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
In healthy women, early menopause is an event that is associated with the exacerbation of several risk factors of cardiovascular and skeletal disease. The occurrence of an early menopause may have even greater impact in women with type 1 diabetes mellitus (DM-1). A small number of studies has demonstrated that DM-1 patients experience cycle irregularity and menopause at a younger age compared to controls. In addition, initial studies have suggested that also in regular cycling DM-1 women a decreased ovarian reserve status for age is present. The explanation for this early decay in ovarian reserve in DM-1 patients remains unknown. Next to auto immunity, vascular factors may be possible contributors to accelerated ovarian ageing in DM-1 patients.

Confirmation of more accelerated ovarian ageing in DM-1 women is urgently needed in view of the added risk factors outlined above. Also, the mechanisms behind the advanced ovarian ageing, with focus on vascular factors, may shed new light on our understanding of the ovarian ageing process per se.

ELIGIBILITY:
Inclusion Criteria:

* Patients: females diagnosed with type 1 diabetes mellitus
* Controls: healthy age-matched female controls

Exclusion Criteria:

* Induced menopause: surgical (premenopausal hysterectomy and/or bilateral ovariectomy), chemo- or radiation therapy, ovarian surgery and irregular menstrual cycles.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part I: Premenopausal women diagnosed with DM-1 older than 18 years and registered at the department for Endocrinology of in several Dutch hospitals.
  Reference group: the Scheffer, Van Rooij, De Vet (SRV) cohort of normal fertile Caucasian women (n=250), recruited in the period of 1990 till 2000.
  For the substudy concerning EPCs will we recruite a control group of 20 healthy female age-matched controls. We will recruite these women within the UMC Utrecht due to logistic reasons.
  Part II: Postmenopausal women diagnosed with DM-1 and registered at the department for Endocrinology of several Dutch hospitals. Reference group:a selection of women from the Prospect-EPIC cohort, who had experienced natural menopause
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
OVADIA 1: serum AMH level | Blood withdrawel once at screening
OVADIA 2: Age at menopause | Assesed once in questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frank Broekmans, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] de Kat AC, Gremmels H, Verhaar MC, Broekmans FJ, Yarde F. Early Vascular Damage in Young Women with DM-1 and Its Relation to Anti-Mullerian Hormone: A Cross-Sectional Study. Int J Endocrinol. 2016;2016:1487051. doi: 10.1155/2016/1487051. Epub 2016 Aug 29. PMID 27651793
- [Derived] Yarde F, van der Schouw YT, de Valk HW, Franx A, Eijkemans MJ, Spiering W, Broekmans FJ; OVADIA study group. Age at menopause in women with type 1 diabetes mellitus: the OVADIA study. Hum Reprod. 2015 Feb;30(2):441-6. doi: 10.1093/humrep/deu327. Epub 2014 Dec 1. PMID 25452435